CLINICAL TRIAL: NCT04744441
Title: Mortality Risk Estimation in Acute Calculous Cholecystitis: Beyond the Tokyo Guidelines
Acronym: ACME
Status: Completed | Type: Observational
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Ana María González Castillo, Principal Investigator, Hospital del Mar
Other Study IDs: Mortality Estimation in ACC
Record Dates: First submitted 2021-01-25; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Acute Calculous Cholecystitis
Keywords: Emergent Cholecystectomy; Mortality in acute Cholecystitis; High Risk Patient; Morbidity in Acute Cholecystitis; Risk Factors in Acute Cholecystitis; Unfit for Surgery; Acute Cholecystitis; Acute Calculous Cholecystitis
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Cholecystectomy; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: CHOLECYSTECTOMY — Surgical treatment
  Other Names: Surgical Treatment
Procedure: PERCUTANEOUS CHOLECYSTOSTOMY — Patients treated with a percutaneous cholecystostomy
  Other Names: Non-Surgical Treatment
Procedure: EXCLUSIVE ANTIBIOTICS — Patients that are treated only with i.v. antibiotics
  Other Names: Non-Surgical Treatment

SUMMARY:
Acute calculous cholecystitis (ACC) is the second most frequent surgical condition in emergency departments, the complication rate of ACC is 20-55%, and the mortality rate is 0.5-15% in recent series. The Tokyo Guidelines (TG) advocate for different initial treatments of ACC with no clear evidence that all patients will benefit from them.

The objective of the study is to identify the risk factors for mortality in ACC and compare them with TG classification.

It is a retrospective cohort study conducted from January 2011 to December 2016 in a single center with a dedicated surgical emergency unit in a Metropolitan University Hospital in Barcelona, Spain. The analysis of the data was finished in March 2020.

The study candidates comprised 963 consecutive patients with a diagnosis of ACC according to the TG18 and/or received a diagnosis of ACC in the Pathology report in those that an emergent cholecystectomy was performed.

The study case definition was a 'Pure Acute Cholecystitis' (pure ACC); therefore, patients with any other concomitant diagnosis potentially influencing outcome (Postoperative cholecystitis, Acute Cholangitis, Acute Pancreatitis, Incidental Cholecystectomy, Acalculous Cholecystitis, Chronic Cholecystitis/Persistent Colic, Post-endoscopic retrograde pancreato-cholangiography, or Neoplasia) were excluded from the final analysis.

Variables:

Primary data were available from a prospective database maintained in File Maker v.12 (Mountainview, CA, USA), which included basic demographic data, type of interventions, sex, days of admission, and complications. Every record was completed by browsing the electronic patient record, adding laboratory and microbiology data, as well as antibiotic therapy, duration of procedure, additional procedures, and grade of acute cholecystitis according to the TG18 diagnostic criteria.

Preoperative comorbidities were assessed using the Charlson Comorbidity Index and surgical risk by ASA classification. The type of initial treatment was classified as Surgical Treatment (Cholecystectomy either by laparoscopy or laparotomy) or Non-Surgical Treatment, which was either percutaneous cholecystostomy or intravenous antibiotics alone.

The main outcome measure was the mortality after the diagnostic of ACC. In the patients that were discharged, 30 days after the diagnosis, if the patients was not discharged in 30 days, at any time during the same admission.

Interventions:

All patients received intravenous antibiotic therapy from the moment the diagnosis was formulated, according to a fixed protocol.

Ultrasound-guided cholecystostomy was performed percutaneously with an 8-Fr catheter (SKATER ™, Argon Medical Devices, Rochester, NY, USA) by either transhepatic or transperitoneal insertion, at the discretion of the radiologist.

Laparoscopic Cholecystectomy was performed according to the French technique using 4 trochars. The content of the gallbladder was evacuated by Veress needle puncture when necessary.

Statistical Analysis:

The normal distribution of the quantitative variables was assessed using the Kolmogorov-Smirnov test, which showed that none of the variables were normally distributed; therefore, their values were expressed as median and interquartile ranges. The Mann-Whitney U non-parametric test was used to assess the significance of differences between means.

The association between qualitative variables was assessed with the chi-square test or Fisher's exact test, as required. The increased risk of an event associated with a variable was reported as the odds ratio (OR) and 95% confidence interval (CI).

As this was a retrospective observational study and the treatment groups were markedly asymmetric, we used the propensity score matching method to select and compare two subgroups of patients evenly balanced by severity according to the TG18 criteria and by comorbidity according to the Charlson Comorbidity Index.

A model for predicting mortality was built using binomial logistic regression with stepwise progressive conditional entry and standard baseline conditions for admission and rejection of variables with significant differences in the univariate analysis. The discrimination power of the model was assessed by receiver operating characteristic (ROC) curves and was compared with the DeLong method.

Legal and Ethical considerations This study was approved by the clinical research ethical committee of the Hospital del Mar and was classified as a non-clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* All patients were selected if they had acute cholecystitis according to the Tokyo Guidelines of 2018 (TG18) and/or received a diagnosis of ACC in the Pathology report. The study case definition was a 'Pure Acute Cholecystitis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admited with a diagnostic of Acute Cholecystitis in a dedicated surgical emergency unit, from January 2011 to December 2016, in a Metropolitan University Hospital in Barcelona, Spain.
Sampling Method: Probability Sample
Enrollment: 963 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
To describe the mortality in patients with a diagnostic of Acute Calculous Cholecystitis. | 2011-2016
  The main outcome measure was the number of deaths after the diagnosis of Acute Calculous Cholecystitis.
  In the patients that were discharged: 30 days after the diagnosis. If the patients was not discharged in 30 days, at any time during the same admission.
To describe the causes of death after a diagnostic of Acute Calculous Cholecystitis | 2011-2016
  Every death after a diagnostic of Acute Calculous Cholecystitis was defined as: septic shock, heart failure, respiratory failure and/or complication of a concomitant chronic disease before the diagnostic of pure ACC.

SECONDARY OUTCOMES:
Study of the risk factors for mortality in patients with a diagnostic of Acute Calculous Cholecystitis | 2011-2016
  The association between qualitative variables was assessed with the chi-square test or Fisher's exact test, as required. The increased risk of an event associated with a variable was reported as the odds ratio (OR) and 95% confidence interval (CI).
  * Demographic data (gender, age)
  * Physiological parameters (Temperature, blood pressure, cardiac and respiratory rates)
  * Laboratory test (Bilirubin, Creatinine, Alkaline phosphatase, Gamma-glutamyl-transpherase, Glutamil oxaloacetic transaminase, PT-INR, Lactate, WBC, Partial oxygen pressure, CRP and Platelets)
  * Type of intervention and additional procedures
  * Grade of severity of ACC following the TG18
  * Preoperative comorbidities were assessed using the Charlson Comorbidity Index and surgical risk by ASA classification.
Comparison the mortality of surgical treatment vs. non-surgical treatment | 2011-2016
  As this was a retrospective observational study and the treatment groups were markedly asymmetric, we performed a propensity score matching method to select patients with an equal morbidity according to the Charlson Comorbidity Index and TG18 Classification at the momento of the diagnostic of ACC. Then we classified the complications of each group following the Clavien-Dindo's Classification.

CONTACTS AND LOCATIONS:
Overall Officials: Ana María González-Castillo, M.D., Principal Investigator — Hospital del Mar

IPD SHARING:
Plan to Share IPD: Yes
all primary and secondary variables of anonimyzed individual data set will be provided
Supporting Information: Study Protocol
Time Frame: January 2021 to January 2022
Access Criteria: any researcher

REFERENCES:
- [Derived] Gonzalez-Castillo AM, Sancho-Insenser J, De Miguel-Palacio M, Morera-Casaponsa JR, Membrilla-Fernandez E, Pons-Fragero MJ, Pera-Roman M, Grande-Posa L. Mortality risk estimation in acute calculous cholecystitis: beyond the Tokyo Guidelines. World J Emerg Surg. 2021 May 11;16(1):24. doi: 10.1186/s13017-021-00368-x. PMID 33975601